CLINICAL TRIAL: NCT00352027
Title: Stanford V Chemotherapy With Low-Dose Tailored-Field Radiation Therapy for Intermediate Risk Pediatric Hodgkin Lymphoma
Brief Title: Chemotherapy With Low-Dose Radiation for Pediatric Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOD05; NCI-2011-01253 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Vinblastine; Mechlorethamine; Cyclophosphamide; Nitrogen Mustard Compounds; Vincristine; Bleomycin; Etoposide; Prednisone; Granulocyte Colony-Stimulating Factor; Filgrastim; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Participants receive 12 weeks of Stanford V chemotherapy which includes Adriamycin®, Vinblastine, Nitrogen Mustard (or Cyclophosphamide), Vincristine, Bleomycin, Etoposide, Prednisone, and G-CSF. After completion of 12 weeks of Stanford V chemotherapy, participants receive radiotherapy.
  Interventions: Drug: Adriamycin®; Drug: Vinblastine; Drug: Nitrogen Mustard; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Bleomycin; Drug: Etoposide; Drug: Prednisone; Biological: G-CSF; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Adriamycin® — Given IV on Day 1 of weeks 1, 3, 5, 7, 9 and 11.
  Other Names: Doxorubicin
Drug: Vinblastine — Given IV, Day 1 of weeks 1, 3, 5, 7, 9 and 11.
  Other Names: Velban®
Drug: Nitrogen Mustard — Given IV, Day 1 of weeks 1, 5 and 9. Cyclophosphamide may be substituted if nitrogen mustard is unavailable.
  Other Names: Mustargen®; Mechlorethamine Hydrochloride
Drug: Cyclophosphamide — May be substituted if nitrogen mustard is unavailable. Given on Day 1 of weeks 1, 5 and 9.
  Other Names: Nitrogen Mustard Derivative
Drug: Vincristine — Given IV on Day 1 of weeks 2, 4, 6, 8, 10 and 12.
  Other Names: Velban®
Drug: Bleomycin — Given IV on Day 1 of weeks 2, 4, 6, 8, 10 and 12.
  Other Names: Blenoxane®
Drug: Etoposide — Given IV on Days 1 and 2 of weeks 1-10.
  Other Names: VP-16; Vepesid®
Drug: Prednisone — Given PO every other day of weeks 1-12.
  Other Names: Synthetic congener of hydrocortisone
Biological: G-CSF — Given subcutaneously days 3-13, 16-26, 29-39, 42-52, 55-65, and 68-78 (as clinically indicated).
  Other Names: Filgrastim; Neupogen®
Procedure: Radiotherapy — Participants receive radiotherapy after completion of 12 weeks of Stanford V chemotherapy.
  Other Names: Radiation therapy

SUMMARY:
The main purpose of this protocol is to estimate the percentage of patients with intermediate risk Hodgkin lymphoma who will survive free of disease (Event-free survival) for three years after treatment with multi-agent chemotherapy (Stanford V) and low-dose, tailored-field radiation therapy. The hypothesis being studied is that this treatment will result in more than 80% of patients being alive and free of disease three years after starting treatment.

DETAILED DESCRIPTION:
Treatment Plan Description:

Adriamycin 25 mg/m2 IV Day 1 of weeks 1, 3, 5, 7, 9, 11

Vinblastine 6 mg/m2 IV Day 1 of weeks 1, 3, 5, 7, 9, 11

Nitrogen Mustard 6mg/m2 IV on Day 1 of weeks 1, 5, and 9

Cyclophosphamide 650 mg/m2 IV Day 1 of weeks 1, 5, 9(when Nitrogen Mustard was not available due to national shortage)

Vincristine 1.4 mg/m2 IV Day 1 of weeks 2, 4, 6, 8, 10, 12

Bleomycin 5 units/m2 IV Day 1 of weeks 2, 4, 6, 8, 10, 12

Etoposide 60 mg/m2 IV Days 1,2 of weeks 3, 7, 11

Prednisone* 40 mg/m2/day divided in 3 doses PO Every other day of weeks 1-12

G-CSF (only as needed in case of severe myelo-suppression requiring treatment delay) 5 mcg/kg SC Days 3-13, 16-26, 29-39, 42-52, 55-65, 68-78 (as clinically indicated)

* Prednisone taper is foreseen for the last 2 weeks of therapy. Patients will be treated with 12 weeks of Stanford V chemotherapy in the schedule outlined above. Patients will then receive radiation therapy after completion of 12 weeks of chemotherapy. The radiation dose to individual nodal sites will be based on response after 8 weeks of chemotherapy: 15 Gy for areas achieving a complete response and 25.5 Gy achieving less than a complete response, or patients with bulky mediastinal mass.

ELIGIBILITY:
Inclusion Criteria:

* Patient is less than or equal to 21 years of age
* Patient has a confirmed diagnosis of previously untreated Hodgkin lymphoma
* Has Ann Arbor stage IB, IIIA, or IA/IIA with extranodal extension, multiple nodal involvement (3 or more sites), or bulky mediastinal adenopathy.

Exclusion Criteria:

* Patients with favorable risk features
* Patients with unfavorable risk features
* Patients who have received prior therapy for Hodgkin lymphoma.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2006-07-20 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Flerlage, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Maine Children's Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between July 2006 and March 2012.
Pre-assignment Details: One participant was determined to be ineligible after enrollment and prior to start of therapy.
Groups:
- Stanford V Chemotherapy: Participants receive 12 weeks of Stanford V chemotherapy:
  Adriamycin, IV, Day 1 of weeks 1, 3, 5, 7, 9 and 11 Vinblastine, IV, Day 1 of weeks 1, 3, 5, 7, 9, 11 Nitrogen Mustard (or Cyclophosphamide), IV, Day 1 of weeks 1, 5, 9 Vincristine, IV, Day 1 of weeks 2, 4, 6, 8, 10, 12 Bleomycin, IV, Day 1 of weeks 2, 4, 6, 8, 10, 12 Etoposide, IV, Days 1, 2 of weeks 1-10 Prednisone, PO, every other day of weeks 1-12 G-CSF, SC, days 3-13, 16-26, 29-39, 42-52, 55-65, 68-78 (as clinically indicated)
  After completion of 12 weeks of Stanford V chemotherapy, participants receive radiotherapy.
Period: Overall Study
Arm/Group | Stanford V Chemotherapy
Started | 80
Completed | 77
Not Completed | 3
Not completed — Progressive disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.10 (3.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 34
Participating Site Location [Number; unit: participants]
  Dana Farber Cancer Institute, Boston, MA | 21
  Main Medical Center, Portland, ME | 2
  Massachusetts General Hospital, Boston, MA | 1
  Rady Children's Hospital, San Diego, CA | 1
  St. Jude Children's Research Hospital, Memphis, TN | 33
  Stanford University Medical Center, Palo Alto, CA | 22

OUTCOME MEASURES:

1. Primary Outcome: 3-year Event-Free Survival Probability
Description: The survival probability for the time interval from treatment start to the time of the first failure (disease recurrence, second malignancy or death) within a 3-year time frame.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
probability | 0.887 [0.821 to 0.959]
Statistical Analysis 1: Comparison: Stanford V Chemotherapy; The association of age with EFS was compared. P values from Score test were computed for the statistical significance; Test type: Superiority or Other; p = 0.9970, Cox Model

2. Secondary Outcome: Disease Failure Rate Within Radiation Fields
Description: Defined as disease that recurs in the initially involved nodal region within the field of irradiation. The disease failure rate within the radiation fields will be estimated with a 95% confidence interval using appropriate methods (e.g., estimate cumulative incidence in the presence of competing risks).
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
proportion of participants | 0.1125 [0.05591 to 0.2076]

3. Secondary Outcome: Local and Distant Failure for Children Treated With Tailored-field Radiation
Description: The cumulative incidence of local and distant failure will be estimated. Effect of competing risks will be taken into account. Local failure is defined as in-field, and distant failure is defined as out-of-field.
Time Frame: from first enrollment date up to 3 years follow-up
Measure: Number (95% Confidence Interval); unit: probability that the event occurs
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
probability that the event occurs
  Cumulative incidence of distant failure at 3 years | 0.0375 [0.0099 to 0.0967]
  Cumulative incidence of local failure at 3 years | 0.1127 [0.0550 to 0.1932]

4. Secondary Outcome: Prognostic Factors for Treatment Failure: Age
Description: Age was examined for the association with event-free survival (EFS) which was defined as the interval between date on study and date of relapse/disease progression, second malignant tumor, death, or last contact, whichever came first. Given only 11 events, the investigators used univariate Cox model with Score test to compute the p value for the statistical significance.
Time Frame: 5.5 (years) median follow-up with minimum 0.3 to maximum 9.4 years follow-up
Measure: Number; unit: events
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
events | 11
Statistical Analysis 1: Comparison: Stanford V Chemotherapy; Test type: Superiority or Other; p = 0.9970, Cox Model

5. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.4.0: Total Score
Description: Patient QOL will be measured at multiple time points to assess the patient's functioning.
  Instrument interpretation: PedsQL v.4.0, higher scores indicate better HRQOL with a range of 0-100.
Time Frame: At Diagnosis (T1), completion of 2 cycles of chemotherapy (T2), completion of 4 cycles of chemotherapy (T3), completion of radiation (T4), and 3-6 months (T5) after the completion of therapy
Population: Each institution made the decision whether to complete the QoL objective. For each time point, a participant and parent proxy completed the QoL questions. Adult participants of majority age did not have a parent proxy.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-therapy: Evaluation completed prior to the start of treatment.
- Week 8: Evaluation completed following 2 courses of therapy, approximately week 8 after start.
- Week 12: Evaluation completed following 4 courses of therapy, approximately week 16 after start.
- After Radiation: Evaluation completed following radiation therapy.
- Off-therapy: Evaluation completed approximately 3-6 months following completion of therapy.
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 58 | 58 | 54 | 38 | 51
units on a scale | 80.9 (12.7) | 74.4 (16.5) | 75.3 (17.8) | 83.1 (14.6) | 84.5 (16.6)

6. Secondary Outcome: Patient Quality of Life (QoL), PedsQl v.4.0: Physical Functioning
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 61 | 60 | 57 | 40 | 54
units on a scale | 83.2 (17.1) | 68.4 (23.1) | 69.1 (24.6) | 80.8 (17.1) | 85.2 (15.6)

7. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.4.0: Psychosocial Health
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 59 | 58 | 54 | 38 | 51
units on a scale | 79.3 (13) | 77.6 (15.4) | 78.6 (16.8) | 84.3 (15.1) | 84.3 (17.9)

8. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.4.0: Emotional Functioning
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 61 | 60 | 57 | 40 | 54
units on a scale | 72.6 (18.0) | 75.3 (19.3) | 75.7 (20.8) | 84.5 (17.8) | 81.6 (24.1)

9. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.4.0:Social Functioning
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 62 | 60 | 57 | 40 | 54
units on a scale | 90.9 (11.1) | 88.6 (13.0) | 88.0 (15.6) | 90.1 (12.5) | 91.1 (13.6)

10. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.4.0: School Functioning
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 60 | 58 | 54 | 38 | 51
units on a scale | 73.1 (18.8) | 69.5 (21.8) | 72.6 (22.2) | 78.4 (20.6) | 81.3 (21.6)

11. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Total Score
Description: Patient QOL will be measured at multiple time points to assess the patient's functioning.
  Instrument interpretation: PedsQL v.3.0, higher scores indicate lower problems with a range of 0-100.
Time Frame: At completion of 2 cycles of chemotherapy (T2), completion of 4 cycles of chemotherapy (T3), completion of radiation (T4), and 3-6 months (T5) after the completion of therapy
Population: Pre-therapy data for PedsQL v.3.0 (symptoms) was not collected, because participants had not started chemotherapy. Each institution made the decision whether to complete the QoL objective. For each time point, a participant and parent proxy completed the QoL questions. Adult participants of majority age did not have a parent proxy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 60 | 57 | 37 | 53
units on a scale |  | 74.1 (15.3) | 74.2 (16.8) | 81.7 (14.6) | 83.5 (17.2)

12. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Pain and Hurt
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 41 | 55
units on a scale |  | 63.9 (25.4) | 71.5 (24.6) | 79.9 (25.1) | 88.0 (17.8)

13. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Nausea
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 41 | 55
units on a scale |  | 62.7 (24.0) | 60.1 (23.5) | 76.7 (20.9) | 81.6 (23.1)

14. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Procedural Anxiety
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 60 | 57 | 40 | 54
units on a scale |  | 71.8 (29.0) | 70.9 (32.6) | 68.1 (37.3) | 80.1 (25.9)

15. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Treatment Anxiety
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 41 | 54
units on a scale |  | 89.2 (15.5) | 82 (22.5) | 89.4 (16.6) | 87.3 (19.1)

16. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Worry
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 41 | 54
units on a scale |  | 71.2 (22.5) | 72.2 (24.7) | 74.5 (27.2) | 76.0 (25.0)

17. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Cognitive Problems
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 41 | 55
units on a scale |  | 79.1 (19.4) | 78.2 (21.4) | 87.0 (17.3) | 82.0 (23.2)

18. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Perceived Physical Appearance
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 38 | 54
units on a scale |  | 77.6 (22.1) | 81.3 (22.6) | 81.4 (22.4) | 84.7 (22.9)

19. Secondary Outcome: Patient Quality of Life (QoL), PedsQL v.3.0: Communication
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 61 | 57 | 39 | 54
units on a scale |  | 80.7 (19.9) | 83.0 (22.5) | 87.2 (22.8) | 89.0 (19.3)

20. Secondary Outcome: Patient Quality of Life (QoL), Symptom Distress Scale
Description: The patient's degree of discomfort from specific treatment-related symptoms across multiple time points.
  Instrument interpretation: SDS, higher scores indicate higher overall symptom distress with a range of 10-50.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 57 | 59 | 52 | 40 | 50
units on a scale | 17.3 (6.5) | 19.6 (6.6) | 18.1 (6.1) | 15.1 (4.8) | 14.3 (5.3)

21. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.4.0: Total Score
Description: Parent's assessment of child's functioning over multiple time points. Instrument interpretation: PedsQL v.4.0, higher scores indicate better HRQOL with a range of 0-100.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 61 | 52 | 50 | 36 | 47
units on a scale | 77.6 (16.7) | 69.1 (17.9) | 72.3 (18.5) | 77.8 (16.3) | 83.5 (16.4)

22. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.4.0: Physical Functioning
Description: as for outcome 21
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 64 | 58 | 56 | 40 | 49
units on a scale | 79.8 (20.7) | 65.3 (23.2) | 67.3 (25.2) | 73.6 (21.3) | 84.6 (18.6)

23. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.4.0: Psychosocial Health
Description: as for outcome 21
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 61 | 52 | 50 | 36 | 47
units on a scale | 76.2 (16.8) | 71.0 (16.7) | 74.1 (17.9) | 79.0 (16.1) | 88.0 (17.0)

24. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.4.0: Emotional Functioning
Description: as for outcome 21
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 64 | 58 | 56 | 40 | 49
units on a scale | 67.7 (20.4) | 65.4 (18.4) | 68.1 (23.7) | 73.0 (20.1) | 82.0 (18.9)

25. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.4.0: Social Functioning
Description: as for outcome 21
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 64 | 58 | 56 | 40 | 49
units on a scale | 86.1 (18.6) | 83.0 (16.0) | 80.7 (18.5) | 85.1 (16.3) | 89.1 (16.8)

26. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.4.0: School Functioning
Description: as for outcome 21
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 61 | 52 | 50 | 36 | 47
units on a scale | 74.4 (20.6) | 62.8 (25.0) | 70.8 (22.7) | 75.6 (20.8) | 78.9 (21.2)

27. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Total Score
Description: Parent's assessment of child's functioning over multiple time points. Instrument interpretation: PedsQL v.3.0, higher scores indicate lower problems with a range of 0-100.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 56 | 55 | 37 | 48
units on a scale |  | 71.7 (16.7) | 69.3 (19.0) | 74.5 (17.7) | 80.0 (16.4)

28. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Pain and Hurt
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 58 | 56 | 40 | 49
units on a scale |  | 61.2 (24.3) | 61.8 (30.5) | 73.1 (25.9) | 82.7 (23.4)

29. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Nausea
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 58 | 57 | 39 | 48
units on a scale |  | 61.2 (24.4) | 57.4 (29.2) | 72.2 (26.6) | 83.2 (22.6)

30. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Procedural Anxiety
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 58 | 55 | 40 | 49
units on a scale |  | 70.0 (32.1) | 60.0 (35.0) | 63.1 (36.6) | 73.8 (31.7)

31. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Treatment Anxiety
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 57 | 56 | 40 | 49
units on a scale |  | 81.9 (21.8) | 72.6 (28.4) | 78.5 (26.8) | 81.8 (20.8)

32. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Worry
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 58 | 56 | 40 | 49
units on a scale |  | 70 (24.5) | 69.2 (25.3) | 71.9 (24.1) | 78.7 (19.4)

33. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Cognitive Problems
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 57 | 55 | 40 | 49
units on a scale |  | 77.6 (21.8) | 79.5 (20.4) | 78.6 (21.8) | 79.9 (23.4)

34. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Perceived Physical Appearance
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 58 | 56 | 38 | 50
units on a scale |  | 74.9 (22.9) | 72.2 (21.9) | 73.7 (24.2) | 76.3 (24.4)

35. Secondary Outcome: Parent Proxy Quality of Life (QoL), PedsQL v.3.0: Communication
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-therapy | Week 8 | Week 12 | After Radiation | Off-therapy
Number analyzed (Participants) | 0 | 58 | 56 | 38 | 50
units on a scale |  | 79.2 (25.9) | 80.4 (24.9) | 80.3 (22.6) | 84.3 (20.3)

36. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.4.0: Total Score
Description: Assess and compare the patient reported and parent proxy quality of life across multiple time points. Reported mean differences were calculated as parent score minus patient score.
  Instrument interpretation: PedsQL v.4.0, higher scores indicate better HRQOL with a range of 0-100. Reported mean differences were calculated as: parent score - patient score.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Parent and Patient Scores at Pre-therapy: Evaluation completed prior to the start of treatment.
- Parent and Patient Scores at Week 8: Evaluation completed following 2 courses of therapy, approximately week 8 after start.
- Parent and Patient Scores at Week 12: Evaluation completed following 4 courses of therapy, approximately week 16 after start.
- Parent and Patient Scores at After Radiation: Evaluation completed following radiation therapy.
- Parent and Patient Scores at Off-therapy: Evaluation completed approximately 3-6 months following completion of therapy.
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 57 | 50 | 49 | 34 | 47
units on a scale | -2.9 (13.3) | -4.8 (13.8) | -4.8 (14.7) | -5 (10.7) | -2.9 (14.8)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Pre-therapy; Test type: Superiority or Other; p = 0.265, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.057, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.079, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.025, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 5: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.680, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

37. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.4.0: Physical Functioning
Description: as for outcome 36
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 60 | 56 | 55 | 37 | 49
units on a scale | -2.9 (16.4) | -2.3 (16.9) | -1.9 (23.3) | -5.4 (15.8) | -2 (19.1)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Pre-therapy; Test type: Superiority or Other; p = 0.563, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.563, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.563, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.184, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 5: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.563, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

38. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.4.0: Psychosocial Health
Description: as for outcome 36
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 58 | 50 | 49 | 34 | 47
units on a scale | -2.8 (14.4) | -6.4 (14.4) | -6.3 (13.2) | -5.6 (11.2) | -3.3 (14.2)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Pre-therapy; Test type: Superiority or Other; p = 0.319, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.010, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.002, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.015, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 5: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.588, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

39. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.4.0: Emotional Functioning
Description: as for outcome 36
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 60 | 56 | 55 | 37 | 49
units on a scale | -4.9 (18.8) | -9.4 (17.9) | -8.0 (14.2) | -10.8 (14.3) | -1.7 (18.8)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Pre-therapy; Test type: Superiority or Other; p = 0.071, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p < 0.001, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 5: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.707, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

40. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.4.0: Social Functioning
Description: as for outcome 36
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 61 | 56 | 55 | 37 | 49
units on a scale | -5.3 (16.5) | -5.7 (15.3) | -7.4 (17.7) | -5.0 (12.6) | -3.3 (16.4)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Pre-therapy; Test type: Superiority or Other; p = 0.042, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.025, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.013, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.027, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 5: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.243, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

41. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.4.0: School Functioning
Description: as for outcome 36
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 59 | 50 | 49 | 34 | 47
units on a scale | 1.3 (17.0) | -5.3 (19.5) | -4.1 (21.0) | -3.4 (16.7) | -4.3 (16.4)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Pre-therapy; Test type: Superiority or Other; p = 0.546, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.242, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.372, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.503, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 5: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.372, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

42. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Total Score
Description: Assess and compare the patient reported and parent proxy quality of life across multiple time points. Reported mean differences were calculated as parent score minus patient score.
  Instrument interpretation: PedsQL v.3.0, higher scores indicate lower problems with a range of 0-100. Reported mean differences were calculated as: parent score - patient score.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 53 | 54 | 33 | 46
units on a scale |  | -1.5 (13) | -5.2 (13.8) | -4.5 (12.5) | -5 (16.8)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.558, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.039, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.162, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.162, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

43. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Pain and Hurt
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 56 | 55 | 38 | 49
units on a scale |  | -2.0 (16.5) | -9.5 (23.6) | -5.6 (23.4) | -5.4 (19.8)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.381, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.006, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.277, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.134, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

44. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Nausea
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 56 | 55 | 37 | 48
units on a scale |  | -1.2 (15.8) | -3.4 (21.9) | -3.0 (22.4) | -1.1 (22.2)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.629, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.629, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.629, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.858, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

45. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Procedural Anxiety
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 55 | 54 | 38 | 48
units on a scale |  | -0.2 (28.1) | -9.3 (29.9) | -2.2 (32.7) | -8.7 (27.7)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.744, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.075, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.512, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.088, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

46. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Treatment Anxiety
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 55 | 55 | 38 | 48
units on a scale |  | -6.1 (21.9) | -8.8 (26.4) | -7.9 (23.7) | -6.6 (26.7)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.078, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.041, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.078, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.078, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

47. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Worry
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 56 | 55 | 38 | 48
units on a scale |  | -0.7 (21.7) | -3.9 (26.5) | -2.7 (20.4) | -0.5 (19.9)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.739, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.739, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.739, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.739, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

48. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Cognitive Problems
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 55 | 54 | 38 | 49
units on a scale |  | -1.0 (20.7) | 0.14 (19) | -8.0 (19) | -4.0 (20)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.933, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.933, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.051, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.0779, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

49. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Perceived Physical Appearance
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 56 | 55 | 34 | 49
units on a scale |  | -2.5 (21.0) | -9.5 (22.5) | -5.9 (25.7) | -9.3 (20.5)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.415, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.005, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.245, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.005, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

50. Secondary Outcome: Correlation of Agreement Between Patient QoL and Parent Proxy QoL at Multiple Time Points, PedsQL v.3.0: Communication
Description: as for outcome 42
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent and Patient Scores at Pre-therapy | Parent and Patient Scores at Week 8 | Parent and Patient Scores at Week 12 | Parent and Patient Scores at After Radiation | Parent and Patient Scores at Off-therapy
Number analyzed (Participants) | 0 | 56 | 55 | 35 | 49
units on a scale |  | -0.3 (26.4) | -3.6 (25.2) | -7.4 (25.5) | -6.3 (21.1)
Statistical Analysis 1: Comparison: Parent and Patient Scores at Week 8; Test type: Superiority or Other; p = 0.814, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 2: Comparison: Parent and Patient Scores at Week 12; Test type: Superiority or Other; p = 0.553, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 3: Comparison: Parent and Patient Scores at After Radiation; Test type: Superiority or Other; p = 0.173, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method
Statistical Analysis 4: Comparison: Parent and Patient Scores at Off-therapy; Test type: Superiority or Other; p = 0.122, Wilcoxon Signed Rank Test — P-values are shown after correction for multiple testing using the False Discovery Rate Method

51. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.4.0: Total Score
Description: Relationship between quality of life and symptom distress instruments aggregated across multiple time points [At diagnosis (T1), completion of 2 cycles of chemotherapy (T2), completion of 4 cycles of chemotherapy (T3), completion of radiation (T4), and 3-6 months (T5) after the completion of therapy]. Generalized estimating equations (GEE) were used to examine the association between symptoms distress and QoL scores.
  Instrument interpretation: PedsQL v.4.0, higher scores indicate better HRQOL with a range of 0-100. SDS, higher scores indicate higher overall symptom distress with a range of 10-50.
Time Frame: 6 months after the completion of therapy
Population: Each institution made the decision whether to complete the QoL objective. For each time point, a participant completed the QoL and symptom distress questions.
Measure: Number (95% Confidence Interval); unit: beta coefficient
Groups:
- QoL Participants: All participants who completed the required questionnaires during at least one time point for evaluating this outcome.
Arm/Group | QoL Participants
Number analyzed (Participants) | 72
beta coefficient | -1.46 [-1.64 to -1.27]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

52. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.4.0: Physical Functioning
Description: as for outcome 51
Time Frame: 6 months after the completion of therapy
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 72
beta coefficient | -1.9 [-2.27 to -1.54]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generallized Estimating Equations (GEE)

53. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.4.0: Psychosocial Health
Description: as for outcome 51
Time Frame: 6 months after the completion of therapy
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 72
beta coefficient | -0.92 [-1.26 to -0.58]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generallized Estimating Equations (GEE)

54. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.4.0: Emotional Functioning
Description: as for outcome 51
Time Frame: 6 months after the completion of therapy
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 72
beta coefficient | -1.56 [-1.95 to -1.16]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generallized Estimating Equations (GEE)

55. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.4.0: Social Functioning
Description: as for outcome 51
Time Frame: 6 months after the completion of therapy
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 72
beta coefficient | -0.79 [-0.98 to -0.59]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generallized Estimating Equations (GEE)

56. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.4.0: School Functioning
Description: as for outcome 51
Time Frame: 6 months after the completion of therapy
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 72
beta coefficient | -1.21 [-1.7 to -0.72]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generallized Estimating Equations (GEE)

57. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Total Score
Description: Relationship between quality of life and symptom distress across multiple time points [completion of 2 cycles of chemotherapy (T2), completion of 4 cycles of chemotherapy (T3), completion of radiation (T4), and 3-6 months (T5) after the completion of therapy]. Generalized estimating equations (GEE) were used to examine the association between symptoms distress and QoL scores.
  Instrument interpretation: PedsQL v.3.0, higher scores indicate better HRQOL with a range of 0-100. SDS, higher scores indicate higher overall symptom distress with a range of 10-50.
Time Frame: 6 months after the completion of therapy
Population: Pre-therapy data for PedsQL v.3.0 (symptoms) was not collected, because participants had not started chemotherapy. Each institution made the decision whether to complete the QoL objective. For each time point, a participant completed the QoL and symptom distress questions.
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -1.41 [-1.71 to -1.11]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

58. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Pain and Hurt
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -2.52 [-3.02 to -2.02]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

59. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Nausea
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -2.31 [-2.85 to -1.77]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

60. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Procedural Anxiety
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -0.87 [-1.49 to -0.26]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p = 0.005, Generalized Estimating Equations (GEE)

61. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Treatment Anxiety
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -0.96 [-1.43 to -0.50]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

62. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Worry
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -1.06 [-1.48 to -0.65]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

63. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Cognitive Problems
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -1.46 [-1.87 to -1.04]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

64. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Perceived Physical Appearance
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -1.20 [-1.68 to -0.72]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

65. Secondary Outcome: Association Between Patient-Reported QoL and Symptom Distress, PedsQL v.3.0: Communication
Description: as for outcome 57
Time Frame: 6 months after the completion of therapy
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: beta coefficient
Arm/Group | QoL Participants
Number analyzed (Participants) | 67
beta coefficient | -1.35 [-1.74 to -0.96]
Statistical Analysis 1: Comparison: QoL Participants; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations (GEE)

66. Secondary Outcome: 3-year Event-free Survival (EFS) Probability
Description: Comparison of thee-year EFS probability along with the whole EFS distributions of intermediate risk patients treated with Stanford V chemotherapy low dose tailored-field radiation to those patients on HOD99.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- HOD05 Participants: Current study defined as Intermediate Risk single arm classified as:
  * EITHER Ann Arbor stage IB and IIIA,
  * OR Ann Arbor stage IA or IIA with ANY of the following features: (1) extranodal extension of disease lesion(s), (2) 3 or more nodal sites involved, (3) Bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph).
  Participants receive 12 weeks of Stanford V chemotherapy:
  Adriamycin, IV, Day 1 of weeks 1, 3, 5, 7, 9 and 11 Vinblastine, IV, Day 1 of weeks 1, 3, 5, 7, 9, 11 Nitrogen Mustard (or Cyclophosphamide), IV, Day 1 of weeks 1, 5, 9 Vincristine, IV, Day 1 of weeks 2, 4, 6, 8, 10, 12 Bleomycin, IV, Day 1 of weeks 2, 4, 6, 8, 10, 12 Etoposide, IV, Days 1, 2 of weeks 1-10 Prednisone, PO, every other day of weeks 1-12 G-CSF, SC, days 3-13, 16-26, 29-39, 42-52, 55-65, 68-78 (as clinically indicated)
  After completion of 12 weeks of Stanford V chemotherapy, participants receive radiotherapy.
- HOD99 Participants: Intermediate Risk participants treated on the earlier HOD99 protocol (NCT00145600) at St. Jude Children's Research Hospital. Intermediate Risk was defined as participants with stage classified as:
  * EITHER Ann Arbor stage IB and IIIA,
  * OR Ann Arbor stage IA or IIA with ANY of the following features: (1) extranodal extension of disease lesion(s), (2) 3 or more nodal sites involved, (3) Bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph).
  Participants received 2 alternating cycles of VAMP/COP chemotherapy (total of 4 cycles of chemotherapy) plus low-dose, involved-field radiotherapy. VAMP chemotherapy includes vinblastine, adriamycin, methotrexate and prednisone. COP chemotherapy includes Cyclophosphamide, Oncovin and Procarbazine.
Arm/Group | HOD05 Participants | HOD99 Participants
Number analyzed (Participants) | 80 | 46
probability | 0.887 [0.821 to 0.959] | 0.844 [0.745 to 0.957]
Statistical Analysis 1: Comparison: HOD05 Participants vs HOD99 Participants; Test type: Superiority or Other; p = 0.908, Log Rank

67. Secondary Outcome: 3-year Overall Survival (OS) Probability
Description: Comparison of the 3-year OS probability along with the whole OS distributions of intermediate risk patients treated with Stanford V chemotherapy low dose tailored-field radiation to those patients on HOD99.
Time Frame: 3-years
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- HOD99 Participants: Intermediate Risk participants treated on the earlier HOD99 protocol (NCT00145600) at St. Jude Children's Research Hospital. Intermediate Risk was defined as participants with stage classified as:
  EITHER Ann Arbor stage IB and IIIA, OR Ann Arbor stage IA or IIA with ANY of the following features: (1) extranodal extension of disease lesion(s), (2) 3 or more nodal sites involved, (3) Bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph).
  Participants received 2 alternating cycles of VAMP/COP chemotherapy (total of 4 cycles of chemotherapy) plus low-dose, involved-field radiotherapy. VAMP chemotherapy includes vinblastine, adriamycin, methotrexate and prednisone. COP chemotherapy includes Cyclophosphamide, Oncovin and Procarbazine.
Arm/Group | HOD05 Participants | HOD99 Participants
Number analyzed (Participants) | 80 | 46
probability | 1.00 [1.00 to 1.00] | 0.978 [0.936 to 1.00]
Statistical Analysis 1: Comparison: HOD05 Participants vs HOD99 Participants; Test type: Superiority or Other; p = 0.178, Log Rank

68. Secondary Outcome: 3-year Local Failure-free Survival Probability
Description: Comparison of the 3-year local failure-free survival probability along with the whole local failure-free survival distributions of intermediate risk patients treated with Stanford V chemotherapy low dose tailored-field radiation to those patients on HOD99.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | HOD05 Participants | HOD99 Participants
Number analyzed (Participants) | 80 | 46
probability | 0.887 [0.821 to 0.959] | 0.932 [0.860 to 1.00]
Statistical Analysis 1: Comparison: HOD05 Participants vs HOD99 Participants; Test type: Superiority or Other; p = 0.411, Log Rank

69. Secondary Outcome: Toxicities With Grade >1
Description: Comparison of the toxicities of intermediate risk patients treated with Stanford V chemotherapy low dose tailored-field radiation (current HOD05 protocol) to those patients on HOD99 (NCT00145600). Grading of toxicities for HOD05 and HOD99 used the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 3 years
Population: Toxicities reported below for the current study (HOD05) include all reported toxicities from a participant's on-study date through 2/17/2016. Toxicities reported below for the HOD99 study include all those reported from a participant's on-study date through their off-study date.
Measure: Number; unit: adverse events
Groups:
- HOD05 - Grade 2; HOD05 - Grade 3; HOD05 - Grade 4; HOD05 - Grade 5: Participants in current study.
- HOD99 - Grade 2; HOD99 - Grade 3; HOD99 - Grade 4; HOD99 - Grade 5: Intermediate Risk participants treated on earlier HOD99 protocol (NCT00145600) at St. Jude Children's Research Hospital.
Arm/Group | HOD05 - Grade 2 | HOD05 - Grade 3 | HOD05 - Grade 4 | HOD05 - Grade 5 | HOD99 - Grade 2 | HOD99 - Grade 3 | HOD99 - Grade 4 | HOD99 - Grade 5
Number analyzed (Participants) | 80 | 80 | 80 | 80 | 46 | 46 | 46 | 46
adverse events
  Alanine transaminase (ALT) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate transaminase (AST) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Allergic reaction/hypersensitivity | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Constipation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Febrile neutropenia | 0 | 7 | 1 | 0 | 0 | 5 | 2 | 0
  Fever (in the absence of neutropenia) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  GGT (gamma-Glutamyltranspeptidase) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin | 0 | 26 | 6 | 0 | 0 | 2 | 0 | 0
  Hypoxia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Ileus, GI (functional obstruction of bowel) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infection with Grade 3 or 4 neutrophils | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
  Infection - Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infection with normal ANC or Grade 1-2 neutrophils | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
  Infection with unknown ANC | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Insomnia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes (total WBC) | 0 | 41 | 15 | 0 | 0 | 19 | 5 | 0
  Lymphopenia | 0 | 22 | 7 | 0 | 0 | 0 | 0 | 0
  Mucositis/stomatitis (functional/symptomatic) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nausea | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Neuropathy: motor | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Neuropathy: sensory | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Neutrophils/granulocytes (ANC/AGC) | 0 | 24 | 32 | 0 | 0 | 9 | 30 | 0
  Pain | 0 | 5 | 0 | 0 | 0 | 1 | 1 | 0
  Phosphate | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
  Potassium | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Syndromes - Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Thrombosis/embolism (vascular access-related) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Thrombosis/thrombus/embolism | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Vomiting | 0 | 2 | 0 | 0 | 1 | 4 | 0 | 0

70. Secondary Outcome: Prognostic Factors for Treatment Failure: Gender
Description: Event-free survival (EFS) was calculated for the 80 eligible patients. EFS was defined as the interval between on study to relapse, second malignant tumor, or last contact (all alive) whichever came first. For those who had multiple relapses, the first one was counted. Given only 11 events, we examined individually age, gender, histology and stage for its association with EFS using Cox model. P values from Score test were computed for the statistical significance.
Time Frame: 3 years follow-up
Measure: Number; unit: events
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
events
  Male | 5
  Female | 6
Statistical Analysis 1: Comparison: Stanford V Chemotherapy; Test type: Superiority or Other; p = 0.4318, Cox Model

71. Secondary Outcome: Prognostic Factors for Treatment Failure: Histology
Description: as for outcome 70
Time Frame: 3 years follow-up
Measure: Number; unit: events
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
events
  Classical, Nodular Sclerosing | 10
  Other | 1
Statistical Analysis 1: Comparison: Stanford V Chemotherapy; Test type: Superiority or Other; p = 0.2199, Cox Model

72. Secondary Outcome: Prognostic Factors for Treatment Failure: Stage
Description: Ann Arbor staging classification was used to stage all patients. Stage was examined (I/II versus III) for the association with event-free survival (EFS), defined as the interval between date on study and of relapse/disease progression, second malignancy, death, or last contact, whichever came first. Given only 11 events, the investigators used univariate Cox model with Score test to compute the p value for the statistical significance. Stage <III showed a better outcome but was not statistically significant.
Time Frame: 5.5 (years) median follow-up with minimum 0.3 to maximum 9.4 years follow-up
Measure: Number; unit: events
Arm/Group | Stanford V Chemotherapy
Number analyzed (Participants) | 80
events
  Stage <III | 8
  Stage ≥III | 3
Statistical Analysis 1: Comparison: Stanford V Chemotherapy; Test type: Superiority or Other; p = 0.8946, Cox Model

73. Secondary Outcome: Describe Toxicities, Particularly the Frequency and Severity of Late Effects of Therapy: (Echocardiogram)
Description: Echocardiograms will be carried out on the patient at 1, 2, 5, and 10 years after therapy. Outcomes will be categorized.
Time Frame: 1, 2, 5, and 10 years post therapy
Population: At each time point, a participant underwent an Echocardiogram (ECHO). Data was unavailable for patients who did not undergo the Echocardiogram at that time point.
Measure: Count of Participants; unit: Participants
Groups:
- Year 1 Off Therapy: Evaluation completed approximately 1 year following completion of therapy.
- Year 2 Off Therapy: Evaluation completed approximately 2 years following completion of therapy.
- Year 5 Off Therapy: Evaluation completed approximately 5 years following completion of therapy.
- Year 10 Off Therapy: Evaluation completed approximately 10 years following completion of therapy.
Arm/Group | Year 1 Off Therapy | Year 2 Off Therapy | Year 5 Off Therapy | Year 10 Off Therapy
Number analyzed (Participants) | 68 | 58 | 38 | 16
Participants
  Normal | 68 | 57 | 36 | 15
  Abnormal | 0 | 1 | 2 | 1

74. Secondary Outcome: Describe Toxicities, Particularly the Frequency and Severity of Late Effects of Therapy: (Electrocardiogram)
Description: Electrocardiograms (EKGs) will be conducted on the patient at 1, 2, 5, and 10 years after therapy. Results will be categorized as either normal or abnormal, determined by the test outcome.
Time Frame: 1, 2, 5, and 10 years post therapy
Population: At each time point, a participant underwent an Electrocardiogram (EKG). Data was unavailable for patients who did not undergo the Electrocardiogram at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Year 1 Off Therapy | Year 2 Off Therapy | Year 5 Off Therapy | Year 10 Off Therapy
Number analyzed (Participants) | 56 | 52 | 28 | 16
Participants
  Normal | 51 | 44 | 24 | 10
  Abnormal | 5 | 8 | 4 | 6

75. Secondary Outcome: Describe Toxicities, Particularly the Frequency and Severity of Late Effects of Therapy: (Pulmonary Function)
Description: Patient pulmonary function will undergo assessment at 1, 2, 5, and 10 years after therapy. Results will be categorized as either normal or abnormal, depending on the test results.
Time Frame: 1, 2, 5, and 10 years post therapy
Population: At each time point, participants who received mediastinal/lung radiation or bleomycin underwent pulmonary function (PFT) assessment. Data was unavailable for patients who did not undergo the pulmonary function test at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Year 1 Off Therapy | Year 2 Off Therapy | Year 5 Off Therapy | Year 10 Off Therapy
Number analyzed (Participants) | 66 | 61 | 36 | 10
Participants
  Normal | 46 | 41 | 25 | 9
  Abnormal | 20 | 20 | 11 | 1

76. Secondary Outcome: Describe Toxicities, Particularly the Frequency and Severity of Late Effects of Therapy: Thyroid (TSH)
Description: For patients that received cervical radiation, TSH laboratory testing will be conducted at 1, 2, 5 and 10 years. TSH results will be categorized as Normal, Hypothyroid, Hyperthyroid, or Thyroid Nodule, depending on the test's findings.
Time Frame: 1, 2, 5, and 10 years post therapy
Population: At each time point, participants who received cervical and upper mediastinal radiation underwent TSH laboratory test. Data was unavailable for patients who did not undergo the TSH test at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Year 1 Off Therapy | Year 2 Off Therapy | Year 5 Off Therapy | Year 10 Off Therapy
Number analyzed (Participants) | 70 | 66 | 46 | 23
Participants
  Normal | 60 | 54 | 37 | 20
  Hypothyroid | 8 | 11 | 8 | 3
  Hyperthyroid | 2 | 1 | 1 | 0
  Thyroid Nodule | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from each participant's on-study date through 4 years after completion of therapy.
Groups:
- Stanford V Chemotherapy: Intermediate risk single arm study defined as
  * EITHER Ann Arbor stage IB and IIIA,
  * OR Ann Arbor stage IA or IIA with ANY of the following features: (1) extranodal extension of disease lesion(s), (2) 3 or more nodal sites involved, (3) Bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph).
  Participants receive 12 weeks of Stanford V chemotherapy:
  Adriamycin, IV, Day 1 of weeks 1, 3, 5, 7, 9 and 11 Vinblastine, IV, Day 1 of weeks 1, 3, 5, 7, 9, 11 Nitrogen Mustard (or Cyclophosphamide), IV, Day 1 of weeks 1, 5, 9 Vincristine, IV, Day 1 of weeks 2, 4, 6, 8, 10, 12 Bleomycin, IV, Day 1 of weeks 2, 4, 6, 8, 10, 12 Etoposide, IV, Days 1, 2 of weeks 1-10 Prednisone, PO, every other day of weeks 1-12 G-CSF, SC, days 3-13, 16-26, 29-39, 42-52, 55-65, 68-78 (as clinically indicated)
  After completion of 12 weeks of Stanford V chemotherapy, participants receive radiotherapy.
Arm/Group | Stanford V Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 69/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanford V Chemotherapy (N=80)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanford V Chemotherapy (N=80)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 56 (111)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 56 (118)
Hemoglobin (Blood and lymphatic system disorders) | 32 (48)
Lymphopenia (Blood and lymphatic system disorders) | 29 (73)
Febrile neutropenia (Infections and infestations) | 8 (11) — Fever of unknown origin without clinically or microbiological documented infection (ANC <1.0 x 10e9/L)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.